CLINICAL TRIAL: NCT00270322
Title: Pain Treatment After Total Knee Replacement - Continuous Epidural Versus Intravenous Patient Controlled Analgesia With Morphine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We believe regional anesth better for TKR,90% patients got epidural. Last year we started spinal morphine one shot, and found it very promissing.
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TKR-1.CTIL
Record Dates: First submitted 2005-12-23; First posted 2005-12-26 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2006-05

CONDITIONS: Pain, Postoperative; Osteoarthritis
Keywords: total knee replacement; orthopedic surgery; post operative analgesia; continuous epidural; patients controlled analgesia; morphine; combined spinal epidural anesthesia; anesthesia; analgesia; epidural marcaine; epidural fentanyl; pain
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis; Agnosia; Pain | interventions — Bupivacaine; Fentanyl; Morphine

INTERVENTIONS:
Drug: Marcaine 0.166% + Fentanyl 3.33 mcg/ml
Drug: Morphine sulphate

SUMMARY:
The study purpose is to compare the effectiveness of different methods for post-operative pain treatment after total knee replacement.

DETAILED DESCRIPTION:
Total knee replacement (TKR) is known to be one of the most painful surgical procedures. Many treatments have been used post TKR: IV opioids, epidural infusions, peripheral nerve blocks. No one method has been recognised as the best one.

In this study we will compare two well established methods of pain treatment:

1. continuous infusion of local anesthetics + opioids into the epidural space,
2. patient controlled analgesia with IV Morphine.

The study design is double blind.

Patients will have a combined spinal-epidural anesthesia for the operation and then will be connected to 2 different pumps, one to the epidural catheter and one to the intravenous catheter, for the first 24 hours post-operatively.

Pain scores, total analgesic medications other than study medications, adverse reactions to study medications, complications and patient satisfaction will be followed by blinded observers and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age: 55 to 85 years
* Osteoarthritis
* Primary unilateral total knee replacement
* American Society of Anesthesiologists (ASA) I-III
* Successful spinal epidural anesthesia for surgery

Exclusion Criteria:

* Any cause for knee replacement other than osteoarthritis
* Total knee revision (re-do)
* Any contraindication for regional anesthesia
* Abnormal coagulation studies
* Thrombocytopenia less than 100,000/cc
* Chronic renal failure (creatinine [cr] < 1.8)
* Neurological disease involving lower extremities
* Major surgery during the last 2 weeks pre-operatively
* Current or past drug or alcohol abuse
* Allergy to study medications
* Post-operative bleeding over 2000 cc/24 hours
* Postdural puncture headache after anesthesia performance

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) (rest/movement) during first 24 hours post-operation
Total dose of rescue analgesics during first 24 hours post-operation

SECONDARY OUTCOMES:
VAS (rest/movement) + total dose rescue analgesics after 24 hours post-operation until discharge
Patient outcome questionnaire
Physiotherapy performance VAS (rest/walking, passive extension, maximal angle, knee flexion/extension)
Adverse reactions, complications

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Edery, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] Williams-Russo P, Sharrock NE, Haas SB, Insall J, Windsor RE, Laskin RS, Ranawat CS, Go G, Ganz SB. Randomized trial of epidural versus general anesthesia: outcomes after primary total knee replacement. Clin Orthop Relat Res. 1996 Oct;(331):199-208. doi: 10.1097/00003086-199610000-00028. PMID 8895639
- [Background] Forst J, Wolff S, Thamm P, Forst R. Pain therapy following joint replacement.A randomized study of patient-controlled analgesia versus conventional pain therapy. Arch Orthop Trauma Surg. 1999;119(5-6):267-70. doi: 10.1007/s004020050407. PMID 10447620
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Singelyn FJ, Deyaert M, Joris D, Pendeville E, Gouverneur JM. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous three-in-one block on postoperative pain and knee rehabilitation after unilateral total knee arthroplasty. Anesth Analg. 1998 Jul;87(1):88-92. doi: 10.1097/00000539-199807000-00019. PMID 9661552
- [Background] Quality improvement guidelines for the treatment of acute pain and cancer pain. American Pain Society Quality of Care Committee. JAMA. 1995 Dec 20;274(23):1874-80. doi: 10.1001/jama.1995.03530230060032. PMID 7500539
- [Background] Foss NB, Kristensen MT, Kristensen BB, Jensen PS, Kehlet H. Effect of postoperative epidural analgesia on rehabilitation and pain after hip fracture surgery: a randomized, double-blind, placebo-controlled trial. Anesthesiology. 2005 Jun;102(6):1197-204. doi: 10.1097/00000542-200506000-00020. PMID 15915033